CLINICAL TRIAL: NCT05120219
Title: A Single-centre, Parallel-cohort, Open-label Study to Assess the Food Effect and Multiple Dose Pharmacokinetic of the HR20033in Healthy Chinese Subjects
Brief Title: A Study to Assess the Effect of Food on HR20033 and Pharmacokinetic After Multiple Dose in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HR20033-102
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: According to the objective, the trial is constituted by two study groups: one is food effect assessment group, and another is multiple dose pharmacokinetic assessment group. There will be 18 (food effect cohort) and 10 (multiple dose pharmacokinetics) volunteers to receive the treatment, and each treatment will be followed by 72 hours of blood sampling for pharmacokinetic assessments, with safety and tolerability.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- food effect cohort A (Experimental)
  Interventions: Drug: FDC tablet
- food effect cohort B (Experimental)
  Interventions: Drug: FDC tablet
- multiple dose pharmacokinetics (Experimental)
  Interventions: Drug: FDC tablet

INTERVENTIONS:
Drug: FDC tablet — single HR20033 FDC tablet fed, take orally on an empty stomach and then after meals
  Arms: food effect cohort A
Drug: FDC tablet — single HR20033 FDC tablet fasted, take orally after meals and then on an empty stomach
  Arms: food effect cohort B
Drug: FDC tablet — single and multiple doses of HR20033 FDC tablet
  Arms: multiple dose pharmacokinetics

SUMMARY:
According to the objective, the trial is constituted by two study groups: one is food effect assessment group, and another is multiple dose pharmacokinetic assessment group.

The primary objective is to (1) assess the effect of a meal (light-fat) on the single-dose PK of SHR3824 and metformin administered in the HR20033 FDC tablet in healthy Chinese subjects; (2) to characterize the single-dose and steady-state PK of SHR3824 and metformin following administration of the HR20033 FDC tablet to healthy subjects in the fed state.

The secondary objective is to assess in healthy Chinese subjects, the safety and tolerability of the SHR3824 and Metformin after single doses (administered in the fed and fasted states) and multiple doses (administered in the fed state) of the HR20033 FDC tablet.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the content, process, and possible adverse reactions of the trial, comply with all study requirements;
2. Male or female subjects aged 18 to 45 (including 18 and 45).
3. Weigh at least 50 kg (for male) and 45 kg (for female), respectively, and have a body mass index (BMI) ≥ 19 and ≤ 26 kg/m2. BMI = weight (kg)/[height (m)]2;
4. The investigator evaluate that the subject meets the standards based on medical history, comprehensive physical examination, laboratory examination, 12-lead electrocardiogram, abdominal B-ultrasound, vital signs, etc.

Exclusion Criteria:

1. Have a birth plan 2 weeks before screening to the end of the follow-up period, or refuse to use medically approved contraceptive measures during this period;
2. Drug abusers or those who test positive for drug abuse screening;
3. Smokers (an average of 5 or more cigarettes per day); or those who quit smoking did not quit for more than 30 days at the time of screening;
4. The average daily alcohol intake in the 1 month before screening exceeds 25 g (for example, 750 mL beer, 250 mL wine or 50 mL low-alcohol liquor); or abstainers have not given up alcohol for more than 30 days at the time of screening;
5. People who have consumed grapefruit or fruit juice products within 2 days before administration, any food or drink containing caffeine (such as coffee, tea, chocolate, cola or other carbonated drinks containing caffeine), purine-rich food or alcohol;
6. The investigator judges that the subject has a medical condition that affects the absorption, distribution, metabolism, and excretion of the drug, or can reduce compliance, or the investigator considers it inappropriate;
7. Hepatitis B surface antigen (HBsAg) positive, or anti-hepatitis C virus (HCV) antibody positive, or human immunodeficiency virus (HIV) antibody positive, or syphilis antibody positive within 1 month before screening or during the screening period;
8. There are any abnormal laboratory test values that are judged by the investigator to be clinically meaningful;
9. The 12-lead electrocardiogram (ECG) is abnormal and has clinical significance;
10. Female subjects are breastfeeding or have a positive serum pregnancy result during the screening period or the test;
11. Any clinical history of serious diseases or diseases or conditions that the investigator believes may affect the test results, including but not limited to the history of circulatory system, endocrine system, nervous system, digestive system, urinary system or blood, immune, mental and metabolic diseases;
12. People with allergies, including those who are clearly allergic to the study drug or any ingredient in the study drug, allergic to any food ingredient or have special dietary requirements, and cannot comply with a unified diet;
13. Those who have undergone any surgery within 3 months before the screening, or who have not recovered after the operation, or who are expected to have surgery or hospitalization plans during the trial period;
14. Those who donated blood (or blood loss) within 3 months before screening and donated blood (or blood loss) ≥400 mL, or received blood transfusion;
15. Those who have participated in clinical trials of any drug or medical device within 3 months before screening;
16. Have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or dietary supplements within 2 weeks before the screening period;
17. Have taken metformin and/or SGLT2 inhibitor drugs such as dapagliflozin, empagliflozin, canagliflozin, and empagliflozin within 1 month before administration.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: Cmax | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: AUC0-t | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: AUC0-inf | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin after single and multiple dose: Cmax | Based on pre-dose, 0.5-72 hours post-dose on day 1 and Day 11, pre-dose on Day 8, Day 9, Day 10 sampling times
Pharmacokinetics parameters of SHR3824 and Metformin after single and multiple dose: AUC0-inf | Based on pre-dose, 0.5-72 hours post-dose on day 1 and Day 11, pre-dose on Day 8, Day 9, Day 10 sampling times
Pharmacokinetics parameters of SHR3824 and Metformin after multiple dose: Cmax，ss | Based on pre-dose, 0.5-72 hours post-dose on day 1 and Day 11, pre-dose on Day 8, Day 9, Day 10 sampling times
Pharmacokinetics parameters of SHR3824 and Metformin after multiple dose: AUCss | Based on pre-dose, 0.5-72 hours post-dose on day 1 and Day 11, pre-dose on Day 8, Day 9, Day 10 sampling times

SECONDARY OUTCOMES:
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: Tmax | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: Vz/F | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: CL/F | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: t1/2 | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin after single and multiple dose: Tmax | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin after single and multiple dose: Ctrough | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin after single and multiple dose: Racc etc | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
The incidence and severity of adverse events/serious adverse events | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided